CLINICAL TRIAL: NCT05194995
Title: A Phase Ib/II Trial of JAB-21822 in Combination With Cetuximab in Patients With Advanced Colorectal Cancer, Small Intestine Cancer and Appendiceal Cancer With KRAS G12C Mutation
Brief Title: JAB-21822 in Combination With Cetuximab in Patients With Advanced CRC and Other Solid Tumors With KRAS G12C Mutation
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Allist Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JAB-21822-1007
Record Dates: First submitted 2021-12-27; First posted 2022-01-18 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-02

CONDITIONS: Advanced Colorectal Cancer; Small Intestinal Cancer; Appendiceal Cancer
MeSH Terms: conditions — Appendiceal Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase 1b Dose Escalation (Experimental): Dose escalation of JAB-21822 to determine maximum tolerated dose of JAB-21822 in combination with cetuximab.
  Interventions: Drug: JAB-21822; Drug: Cetuximab
- Phase 2 Dose Expansion, Cohort 1 (Experimental): Enrollment into the dose expansion cohort is for eligible participants with KRAS P.G12C mutant advanced colorectal cancer.
  Interventions: Drug: JAB-21822; Drug: Cetuximab
- Phase 2 Dose Expansion, Cohort 2 (Experimental): Enrollment into the dose expansion cohort is for eligible participants with KRAS P.G12C mutant advanced small intestinal cancer and advanced appendiceal cancer.
  Interventions: Drug: JAB-21822; Drug: Cetuximab

INTERVENTIONS:
Drug: JAB-21822 — JAB-21822 administered orally as a tablet.
Drug: Cetuximab — Cetuximab administered as an intravenous (IV) infusion.

SUMMARY:
This study is to evaluate the safety, tolerability, pharmacokinetics and antitumor activity of JAB-21822 in combination with cetuximab in patients with advanced colorectal cancer，advanced small intestine cancer and advanced appendiceal cancer with KRAS p.G12C mutation.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and tolerability of JAB-21822 in combination with cetuximab to determine the MTD and RP2D during Dose Escalation phase; then to evaluate preliminary antitumor activity when JAB-21822 is administered in combination with cetuximab during Dose Expansion phase in patients with advanced colorectal cancer，advanced small intestine cancer and advanced appendiceal cancer with KRAS p.G12C mutation.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be able to provide an archived tumor sample
* Histologically or cytologically confirmed advanced colorectal cancer, advanced small intestinal cancer and advanced appendiceal cancer with KRAS p.G12C mutation
* Must have received at least 1 prior standard therapy
* Must have at least 1 measurable lesion per RECIST v1.1
* Must have adequate organ function
* Must be able to swallow and retain orally administered medication

Exclusion Criteria:

* Has brain metastases, except if treated and no evidence of radiographic progression or hemorrhage for at least 28 days
* Active infection requiring systemic treatment within 14 days
* Active HIV, HBV or HCV
* Any severe and/or uncontrolled medical conditions
* LVEF<50% assessed by ECHO
* QT interval >470 msec

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation phase: Number of participants with dose-limiting toxicities (DLTs) | At the end of Cycle 1 (each cycle is 21 days)
  A DLT is defined as the clinically significant treatment related adverse event (TRAE) or abnormal laboratory values assessment during the first 21 days of (Cycle 1) and excludes events that are deemed clearly related to underlying disease, progression, or intercurrent illness.
Dose Expansion phase: Overall response rate (ORR) | Up to 4 years - from baseline to RECIST confirmed Progressive Disease
  ORR is defined as the percentage of participants with complete response (CR) or partial response (PR) per RECIST v 1.1.

SECONDARY OUTCOMES:
Dose Escalation and Dose Expansion phase: Number of participants with adverse events | Up to 4 years
  Patients will be assessed for incidence and severity of adverse events (AEs) according to NCI-CTCAE criteria.
Dose Escalation and Dose Expansion phase: Peak Plasma Concentration (Cmax) | Up to 4 years
  Cmax of JAB-21822 will be measured by using plasma PK samples.
Dose Escalation and Dose Expansion phase: Area under the plasma concentration versus time curve (AUC) | Up to 4 years
  AUC of JAB-21822 will be measured by using plasma PK samples.
Dose Expansion phase: Duration of response ( DOR ) | Up to 4 years
  DOR is defined as the time from the participant's initial objective response (CR or PR) to disease progression per CTCAE v1.1 or death due to any cause, whichever occurs first.
Dose Escalation phase: Overall response rate (ORR) | Up to 4 years
  The percentage of participants with complete response (CR) or partial response (PR) on RECIST v 1.1.
Dose Expansion phase: Disease Control Rate ( DCR ) | Up to 4 years
  DCR is defined as percentage of participants with complete response (CR), partial response (PR), or stable disease(SD) per CTCAE v1.1.
Dose Expansion phase: Progression-free survival (PFS) | Up to 4 years
  PFS is defined as the interval of time between the date of first treatment to the earliest date of disease progression per CTCAE v1.1 or death which occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Shen Lin Master of medicine, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (17):
- China (17):
  - Research site31, Beijing, Beijing Municipality
  - Research site01, Beijing, Beijing Municipality
  - Research site02, Beijing, Beijing Municipality
  - Research site12, Beijing, Beijing Municipality
  - Research site13, Nanning, Guangxi
  - Research site06, Harbin, Heilongjiang
  - Research site05, Zhengzhou, Henan
  - Research site07, Zhengzhou, Henan
  - Research site18, Wuhan, Hubei
  - Research site11, Changsha, Hunan
  - Research site29, Changsha, Hunan
  - Research site09, Nanjing, Jiangsu
  - Research site08, Nanchang, Jiangxi
  - Research site16, Linyi, Shandong
  - Research site28, Shanghai, Shanghai Municipality
  - Research site23, Xi’an, Shanxi
  - Research site19, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Li J, Wang Z, Huang J, Ba Y, Cao B, Luo S, Li W, Bai C, Song Z, Xiong J, Zhu L, An G, Zhang Y, Li Z, Li Y, Gu Y, Hu C, Li X, Huang C, Fu Q, Yin X, Liang X, Zhong D, Shi H, Li X, Li Z, Liu L, Wang F, Liang R, Xia G, Wang Z, Wang-Gillam A, Ding Y, Rao Z, Pan W, Lu S, Sun X, Shen L. Glecirasib with or without cetuximab in previously treated locally advanced or metastatic colorectal cancer with KRASG12C mutation (JAB-21822-1002 and JAB-21822-1007): two open-label, non-randomised phase 1/2 trials. Lancet Gastroenterol Hepatol. 2026 Feb;11(2):110-123. doi: 10.1016/S2468-1253(25)00267-5. Epub 2025 Dec 1. PMID 41344351